CLINICAL TRIAL: NCT03008096
Title: Laparoscopic Sleeve Gastrectomy as Bridge-to-Candidacy for Obese Left-Ventricular Assist Device Patients
Acronym: LSG-BTC-LVAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philipp Angleitner (Other)
Responsible Party: Sponsor-Investigator, Philipp Angleitner, Resident, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSG-BTC-LVAD
Record Dates: First submitted 2016-12-16; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Heart Failure; Obesity
MeSH Terms: conditions — Heart Failure; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Laparoscopic Sleeve Gastrectomy — Routine Laparoscopic Sleeve Gastrectomy is performed on obese patients supported by Left-Ventricular Assist Device in order to reach a Body Mass Index sufficient for heart transplantation listing.
  Other Names: Bariatric Surgery

SUMMARY:
In LVAD (Left-Ventricular Assist Device) patients, evidence is lacking regarding the safety and efficacy of Laparoscopic Sleeve Gastrectomy (LSG) as a means to reach a Body Mass Index (BMI) within listing criteria for heart transplantation. To our knowledge, this is the first prospective study to evaluate laparoscopic sleeve gastrectomy in LVAD patients as bridge-to-candidacy for heart transplantation.

DETAILED DESCRIPTION:
Continuous-flow left-ventricular assist devices are increasingly used for the treatment of acute or chronic end-stage heart failure (Mancini 2015). Three main implantation strategies exist: destination therapy (support until end of life), bridge to transplantation (support until transplantation), and bridge to candidacy (support until transplantation criteria are met). Although LVAD support delivers excellent short-term and long-term results, the current gold standard and last resort of treatment for end-stage heart failure remains orthotopic heart transplantation (Lund 2015).

Obesity increases mortality in heart transplantat recipients and therefore is included in the 2006 transplantation criteria. The heart transplant program of the Medical University of Vienna uses a BMI of 30 kg/m2 as the upper limit to be listed for heart transplantation (Mehra 2016).

Ambulatory patients on CF-LVAD support have a tendency to gain weight because of reduced physical fitness, inability to work, and genetic predisposition. In many cases, binge eating is used as a coping mechanism to alleviate depression and anxiety associated with heart failure and LVAD therapy.

Conservative measures to reduce weight and increase physical fitness fail in many patients. As a result, in many cases these patients remain ineligible for heart transplantation for months or years. For the entire period of ineligibility, they are subject to the constant life-threatening risks of LVAD treatment, most importantly ischemic and hemorrhagic stroke, pump thrombosis, infection, right heart failure, and bleeding episodes in the gastrointestinal tract or other organ systems (Kirklin 2015).

Bariatric surgery has been shown to be superior to conservative measures of weight reduction in morbidly obese patients. Laparoscopic sleeve gastrectomy, one of the most commonly employed bariatric procedures, reduces body weight by a non-malabsorptive mechanism (Colquitt 2014). Gastric volume reduction is achieved by resection along the stomach's greater curvature and creation of a gastric tube, leading to reduced capacity for ingested food, decreased appetite and earlier satiety. In contrast to malabsorptive bariatric procedures, resorption and efficacy of immunosuppressive drugs, an inevitable feature of post-transplant therapy, are only minimally influenced following sleeve gastrectomy. Furthermore, there is less requirement for substitution of trace elements and vitamins, for example Vitamin B12. Due to the fact that the majority of obese LVAD patients are within a BMI range of 30 to 40 kg/m2, the moderate weight loss achieved by sleeve gastrectomy is expected to be sufficient for reaching the eligibility criterion for heart transplantation.

It is unclear, whether laparoscopic sleeve gastrectomy is effective and safe in patients on CF-LVAD. The literature is limited to case reports and retrospective series of up to 4 patients. This is the first prospective series including more than 4 patients with the specific aim to enable obese LVAD supported patients to reach a BMI within listing criteria for heart transplantation by the means of laparoscopic sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients on LVAD-support for end-stage heart failure
* Bridge-to-Candidacy strategy
* BMI > 35kg/m2
* Failure to reach BMI < 30kg/m2 with conservative measures
* Age > 18 years
* Ability to give informed consent

Exclusion Criteria:

- Absolute contraindications to subsequent heart transplantation other than obesity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
BMI (Body-Mass-Index) | 12 months post-LSG
  Patient weight is measured and BMI is calculated at the time of LSG and at 3, 6, and 12 months post-LSG. The rate of patients with successful weight reduction to a BMI lower than 30kg/m2 is calculated.

SECONDARY OUTCOMES:
NYHA (New York Heart Association) Class | 12 months post-LSG
  Patients' NYHA Class (I, II, IIIa, IIIb, IV) is assessed pre-operatively and at 3, 6, and 12 months post-LSG and changes are noted.
6-min Walking Test | 12 months post-LSG
  Patients are performing the 6-min walking test pre-operatively and at 3, 6, and 12 months post-LSG and changes of the distance walked (m) are assessed.
EQ-5D (EuroQol five dimensions) questionnaire | 12 months post-LSG
  Patients are undertaking the EQ-5D quality-of-life questionnaire (mobility, self care, usual activities, pain/discomfort, anxiety/depression, and visual analog scale) pre-operatively and at 3, 6, and 12 months post-LSG to assess changes in the post-operative quality of life.
Work Ability questionnaire | 12 months post-LSG
  Patients are undertaking the Work Ability questionnaire including questions about their current or former occupation pre-operatively and at 3, 6, and 12 months post-LSG to assess changes in occupational issues.
WHOQOL-BREF (World Health Organization Quality of Life) questionnaire | 12 months post-LSG
  Patients are undertaking the WHOQOL-BREF questionnaire including questions regarding their quality of life pre-operatively and at 3, 6, and 12 months post-LSG to assess changes regarding social, emotional, and health-related issues.
LVEF (Left-Ventricular Ejection Fraction) | 12 months post-LSG
  LVEF (%) is going to be measured by echocardiography pre-operatively and at 3, 6, and 12 months post-LSG to investigate changes of cardiac function.
VO2 max (maximum rate of oxygen consumption) | 12 months post-LSG
  Patients are undergoing spiroergometry pre-operatively and at 3, 6, and 12 months post-LSG to investigate changes of cardiac performance.
Severe adverse events | 12 months post-LSG
  Adverse and severe adverse events including death, unplanned hospital readmission, reoperation, major bleeding, cardiac arrhythmia, pericardial fluid collection, device malfunction, hemolysis, hepatic dysfunction, hypertension, major infection, myocardial infarction, neurological dysfunction, psychiatric episodes, renal dysfunction, respiratory failure, right heart failure, arterial non-CNS (central nervous system) thromboembolism, venous thromboembolism, wound dehiscence, gastroesophageal reflux disease, vomiting, gastric anastomotic leak, trocar site infection, trocar site hernia, gastric pouch dilation, and others are assessed in the immediately post-operative phase and at 3, 6, and 12 months post-LSG.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Zimpfer, Priv.-Doz. Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Division of Cardiac Surgery, Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mancini D, Colombo PC. Left Ventricular Assist Devices: A Rapidly Evolving Alternative to Transplant. J Am Coll Cardiol. 2015 Jun 16;65(23):2542-55. doi: 10.1016/j.jacc.2015.04.039. PMID 26065994
- [Background] Lund LH, Edwards LB, Kucheryavaya AY, Benden C, Dipchand AI, Goldfarb S, Levvey BJ, Meiser B, Rossano JW, Yusen RD, Stehlik J. The Registry of the International Society for Heart and Lung Transplantation: Thirty-second Official Adult Heart Transplantation Report--2015; Focus Theme: Early Graft Failure. J Heart Lung Transplant. 2015 Oct;34(10):1244-54. doi: 10.1016/j.healun.2015.08.003. Epub 2015 Aug 28. No abstract available. PMID 26454738
- [Background] Mehra MR, Canter CE, Hannan MM, Semigran MJ, Uber PA, Baran DA, Danziger-Isakov L, Kirklin JK, Kirk R, Kushwaha SS, Lund LH, Potena L, Ross HJ, Taylor DO, Verschuuren EAM, Zuckermann A; International Society for Heart Lung Transplantation (ISHLT) Infectious Diseases, Pediatric and Heart Failure and Transplantation Councils. The 2016 International Society for Heart Lung Transplantation listing criteria for heart transplantation: A 10-year update. J Heart Lung Transplant. 2016 Jan;35(1):1-23. doi: 10.1016/j.healun.2015.10.023. No abstract available. PMID 26776864
- [Background] Kirklin JK, Naftel DC, Pagani FD, Kormos RL, Stevenson LW, Blume ED, Myers SL, Miller MA, Baldwin JT, Young JB. Seventh INTERMACS annual report: 15,000 patients and counting. J Heart Lung Transplant. 2015 Dec;34(12):1495-504. doi: 10.1016/j.healun.2015.10.003. Epub 2015 Oct 8. PMID 26520247
- [Background] Colquitt JL, Pickett K, Loveman E, Frampton GK. Surgery for weight loss in adults. Cochrane Database Syst Rev. 2014 Aug 8;2014(8):CD003641. doi: 10.1002/14651858.CD003641.pub4. PMID 25105982